CLINICAL TRIAL: NCT05072587
Title: Dietary Oxysterols and β-Cell Function Among African Americans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Jennifer Rooke, MD, MPH, Assistant Professor, Morehouse School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MorehouseSM
Record Dates: First submitted 2021-09-24; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes
Keywords: Beta-cell dysfunction oxysterols African Americans
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: This pilot study is a longitudinal prospective randomized clinical trial with two parallel arms. Participants in both arms of the study will receive prepared meals based on ADA dietary guidelines for 12 weeks. One group will be given a plant-based ADA diet that contains no oxysterols (PB-ADAØ). The other group will be given the Standard ADA diet (SADA). The dietary 7-KC content of both diets will be estimated from oxysterol food composition databases. Sample meals from both groups will be analyzed to determine the 7-KC food content and the accuracy of the estimates.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Standard ADA dietary guidelines (SADA) (Active Comparator): Participants in this group will be given prepared meals based on standard ADA dietary guidelines for 12 weeks.
  Interventions: Behavioral: Standard ADA Diet (SADA)
- Group B - Plant Based ADA diet with no oxysterols (PB-ADAØ). (Experimental): Participants in this group will be given prepared meals based on ADA guidelines but with no dietary cholesterol oxides/oxysterols - Plant-based ADA diet
  Interventions: Behavioral: Plant-based diet with no oxysterols

INTERVENTIONS:
Behavioral: Plant-based diet with no oxysterols — This group will be given 3 prepared plant-based meals a day with macronutrient content: 60% of calories from carbohydrates, 15% protein, and 25% fat. Calories: 25 kcal/kg ideal body weight (IBW). The goal is weight maintenance, but weight loss may occur. 1-5% weight loss will be acceptable and not deemed a potential confounder. Participants will be screened for food allergies and intolerances prior to receiving their research diets. All meals will include culturally familiar foods to enhance adherence. The dietary intervention will be conducted over 4 3-month periods (12 months). Meals will be packaged labeled and distributed to participants once per week. Participants will consume their meals at home.
  Other Names: Cholesterol Oxide-free plant-based diet
  Arms: Group B - Plant Based ADA diet with no oxysterols (PB-ADAØ).
Behavioral: Standard ADA Diet (SADA) — This group will be given 3 prepared meals a day with macronutrient content: 60% of calories from carbohydrates, 15% protein, and 25% fat. Calories: 25 kcal/kg ideal body weight (IBW). The goal is weight maintenance, but weight loss may occur. 1-5% weight loss will be acceptable and not deemed a potential confounder. Participants will be screened for food allergies and intolerances prior to receiving their research diets. All meals will include culturally familiar foods to enhance adherence. The dietary intervention will be conducted over 4 3-month periods (12 months). Meals will be packaged labeled and distributed to participants once per week. Participants will consume their meals at home.
  Other Names: ADA Diet
  Arms: Group A - Standard ADA dietary guidelines (SADA)

SUMMARY:
African Americans (AAs) have a higher risk of developing type 2 diabetes than the general population. AAs are also more likely to eat foods that contain cholesterol oxides/oxysterols.

Dietary oxysterols can harm the cells that produce insulin and decrease insulin production.

This pilot study seeks to determine if removing dietary oxysterols with a plant-based diet will improve insulin production and decrease the risk of type 2 diabetes among AAs.

DETAILED DESCRIPTION:
African Americans (AAs) have almost twice the incidence and prevalence of Type 2 diabetes (T2D) compared to the general population. T2D occurs when pancreatic β-cell dysfunction prevents secretion of sufficient insulin to overcome insulin resistance. While the causes of β-cell dysfunction are not fully understood, the role of cytotoxic oxidative stress is well documented. Serum oxysterols are biomarkers of oxidative stress. Oxysterols form endogenously or exogenously when cholesterol in food is exposed to light, heat, and processing. Dietary oxysterols are cytotoxic, they are absorbed and carried in the blood by lipoprotein carriers or circulate freely in serum. 7-Ketocholesterol (7-KC), the most common oxysterol in food and serum is a biomarker of cholesterol oxidation. High serum levels of 7-KC are associated with an increased risk of T2D. AAs who consume Southern dietary pattern foods such as fried and processed meats have a higher consumption of dietary oxysterols than the general population. Our central hypothesis is that the higher consumption of dietary oxysterols among AAs contributes to β-cell dysfunction and higher rates of T2D. The aim of this pilot study is to determine the effect of lowering dietary oxysterols on serum 7-KC and β-cell function among AAs with prediabetes and early T2D (HbA1c 5.7% - 7.0%). The expected outcome is that decreased exposure to dietary oxysterols will decrease serum oxysterols and β-cells oxidative stress which will improve β-cell function and glycemic control. The knowledge gained from this study may lead to improved T2D prevention and treatment strategies that may decrease the burden of T2D in all communities and eliminate the racial disparity among AAs.

ELIGIBILITY:
Inclusion Criteria: Participants must be:

1. HbA1c: 5.7% - 7.0%: This HbA1c range reflects mild to moderate β-cell dysfunction.
2. Self-identified AA: This group has higher rates of T2D than the general population.
3. Adults over18 years old: This age group is at higher risk of T2D.
4. Ability to read, understand and communicate effectively in English: All information about the study and instructions for the study protocol will be in English.
5. Committed to eating the allocated study diet for 12 weeks: This is important to ensure that the study protocol is followed, and the data collected from participants is meaningful/valid.
6. On stable medication dosages for the three months prior to recruitment: This is to avoid bias or confounding with new medications or dosages changes.
7. Able to safely store a week's supply of prepared meals: Participants will receive packages of prepared food that has to stored and last them for the following week.
8. Mentally competent and able to follow the study protocol and provide informed consent
9. Currently eating the Standard American diet: The baseline diet of the participants will be assessed and correlated their baseline serum 7-KC levels and HOMA2 Index of β-cell function.

Exclusion Criteria: Participants cannot:

1. Be pregnant or lactating: Fetuses and breast-feeding infants are a protected vulnerable group. The risk of involving them in research must outweigh the benefits, Hormonal levels and other factors in pregnant and lactating woman may confound study results.
2. Be taking statin medications or any other cholesterol lowering drugs or supplements: These medications may artificially lower serum cholesterol and oxysterol levels.
3. Be currently on a vegan, vegetarian, or any type of plant-based diet for the 3 months prior to recruitment: Participants currently on these diets may not see significant changes on the dietary interventions of the study protocol.
4. Be a current smoker: Smoking is a risk factor for oxidative stress - this could be an effect modifier or a confounding faction for this study.
5. Be on medications or supplements to lower blood glucose or treat diabetes: This will be an effect modifier or confounding factor. We will not know the effect of the dietary intervention if the participants are also on medications for diabetes.
6. Be status post blood transfusion in the previous 3 months: This will interfere with the test for HbA1c levels. This is one of our primary outcomes:
7. Have a hemoglobin or any other blood disorder: This will interfere with the test for HBA1c which measures glycation of hemoglobin in red blood cells.:
8. Be taking biotin supplements: This interferes with the test for fasting C-Peptide.
9. Be on dialysis or have any stage of renal failure: Dialysis patients need special diets and more intense monitoring than is planned for the participants in this study.
10. Have food allergies: Participants will be screened for food allergies. This is to prevent food sensitivities or adverse reactions to the prepared meals in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
The Homeostasis Model Assessment of β-cell function (HOMA-B) Index | 12 Weeks
  The HOMA-B index will be calculated using the HOMA2 Calculator with fasting C-peptide and fasting blood glucose levels. This study will compare the effect of the standard American Diabetes Association (ADA) diet that contains oxysterols and a plant-based ADA diet that does not contain oxysterols on the HOMA-B index of African Americans (AAs) with prediabetes and early diabetes.
Glycated Hemoglobin (HbA1c) | 12 weeksC-peptide levels are elevated in renal failure It is produced in equim C
  HbA1c is a measure of glycemic control. This study will compare the effect of the standard ADA diet that contains oxysterols and a plant-based ADA diet without oxysterols on the HbA1c of AAs with HbA1c levels between 5.7% and 7.0%.
Serum 7-Ketocholesterol (7-KC) | 12 weeks
  7-KC is one of the most abundant oxysterols in food and serum. This study will compare the effect of a standard ADA diet with oxysterols and a plant-based ADA diet without oxysterols on serum 7-KC levels. 7-KC will be measured by tandem liquid chromatography /mass spectrometry at the Emory Lipidomics lab.

SECONDARY OUTCOMES:
The Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) Index | 12 Weeks
  This index will be calculated using the HOMA2 Calculator with fasting insulin and fasting blood glucose levels. The impact of the 2 different study diets on the HOMA-IR will be determined.
Fasting Insulin | 12 weeks
  Insulin is a hormone produced by beta cells in the pancreas, it regulates serum glucose levels. The impact of the 2 different study diets on fasting insulin will be determined.
Fasting C-Peptide | 12 weeks
  C-peptide is a short chain of amino acids that is released as a byproduct of insulin production. It is produced in equimolar amounts as endogenous insulin but excreted at a more constant rate over a longer time. It is a sensitive, clinically validated assessment of of β-cell function. This study will measure the effect of the 2 study diets on fasting C-peptide.
Fasting Blood Glucose | 12 weeks
  Glucose is the main sugar found in blood. Elevated fasting blood glucose is a sign of diabetes. This study will measure the effects of the 2 study diets on fasting blood glucose.
Total cholesterol (TC) | 12 weeks
  TC is a measure of the total amount of cholesterol in blood. This study will determine the effect of the 2 study diets on serum TC levels.
High Density Lipoproteins (HDL) | 12 weeks
  HDL is the lipoprotein carrier that carries cholesterol from the cell to the liver to be excreted. This study will measure the effect of the 2 study diets on serum HDL levels.
Low Density Lipoproteins (LDL) | 12 weeks
  LDL is the liproprotein carrier that carries cholesterol from the liver to the cells of the body. This study will measure the effect of the 2 study diets on serum LDL levels.
Oxided Low Density Lipoproteins (Ox-LDL) | 12 weeks
  Ox-LDL form when LDLs carry cholesterol oxides/oxysterols. Ox-LDLs are cytotoxic and better indicators of cardiovascular risk than native LDL levels. This study will measure the effect of the 2 study diets on serum LDL levels.
Aspartate Amino Transferase (AST) | 12 weeks
  AST is an enzyme that is released from the liver when it is injured. It is an indicator of liver function. This study will measure the effect of the 2 study diets on AST levels.
Alanine Amino Transferase (ALT) | 12 weeks
  ALT is an enzyme that is released from the liver when it is injured. It is an indicator of liver function. This study will measure the effect of the 2 study diets on ALT levels.
Glomerular Filtration Rate (GFR) | 12 weeks
  GFR is an index of kidney function. This study will measure the effect of the 2 study diets on GFR. In addition, it is important to measure kidney function in this study because C-peptide levels are elevated in renal failure
Blood Urea Nitrogen (BUN) | 12 weeks
  BUN is a breakdown product of protein that is cleared from the blood by the kidneys. It is an indicator of kidney function. This study will measure the effect of the 2 study diets on BUN.
Creatinine | 12 weeks
  Creatinine is a by-product of normal muscle breakdown that is cleared from the blood by the kidneys. It is an indicator of kidney function. This study will measure the effect of the 2 study diets on serum creatinine levels.
White Blood Cell (WBC) Count | 12 weeks
  The WBC count is a measure of the number of WBCs the body. WBCs are immune cells and markers of inflammation. This study will measure the effect of the 2 study diets on WBC counts.
Hemoglobin (Hb) | 12 weeks
  Hb is a protein in red blood cells that carries oxygen from the lungs to the body. This study will measure the effect of the 2 study diets on Hb levels. In addition, it is important to know Hb levels because Hb abnormalities affect HbA1c levels.
Platelet Count | 12 weeks
  The platelet count is the number of platelets in blood. Platelets are involved in clotting, which is dysfunctional in diabetes. This study will measure the effect of the 2 study diets on platelet counts.
Calcium | 12 weeks
  This is measure of serum calcium levels. A plant-based diet may cause low calcium levels. This study will measure the effect of the 2 study diets on serum calcium levels.
Vitamin B12 | 12 weeks
  This is a measure of vitamin B-12 levels. People on plant-based diets may have lower vitamin B12 levels. This study will measure the effect of the 2 study diets on vitWBC amin B12 levels.
Blood pressure (BP) | 12 weeks
  BP is the pressure of circulating blood against the walls of blood vessels. It is an indicator of cardiovascular health. It will be measured at baseline, 6-weeks and post intervention. This study will measure the effect of the 2 study diets on BP.
Body composition using the Dual X-ray Absorptiometry (DEXA) Body Composition scan | 12 weeks
  The DEXA scan provides an analysis of body fat, muscle mass and bone density. This study will measure the effect of the 2 study diets on body composition.
Body Mass Index (BMI) | 12 weeks
  BMI is defined as the body weight divided by the square of the body height. This is expressed in units of kg/m². It will be used to classify study particpants according to body mass into underweight, normal, overweight or obese groups. This study will measure the effect of the 2 study diets on BMI.
Waist circumference (WC) | 12 weeks
  WC is the measurement taken around the abdomen at the level of the umbilicus (belly button). This measures abdominal obesity which may be a better indicator of health risk than BMI. This study will measure the effect of the 2 study diets on WC.
World Health Organization (WHO-5) Index of Well Being | 12 weeks
  The WHO-5 Well-Being Index is a short self-reported measure of current mental wellbeing. This study will measure the effect of the 2 study diets on this indicator of well being.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rooke, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Background] Diabetes and African Americans, CDC 2016. Summary Health Statistics: National Health Interview Survey: 2014. US Department of Health and Human Services, Office of Minority Health website. http://www.cdc.gov/nchs/nhis/shs/tables.htm
- [Background] Benoit SR, Hora I, Albright AL, Gregg EW. New directions in incidence and prevalence of diagnosed diabetes in the USA. BMJ Open Diabetes Res Care. 2019 May 28;7(1):e000657. doi: 10.1136/bmjdrc-2019-000657. eCollection 2019. PMID 31245008
- [Background] Staimez LR, Rhee MK, Deng Y, Safo SE, Butler SM, Legvold BT, Jackson SL, Ford CN, Wilson PWF, Long Q, Phillips LS. Retinopathy develops at similar glucose levels but higher HbA1c levels in people with black African ancestry compared to white European ancestry: evidence for the need to individualize HbA1c interpretation. Diabet Med. 2020 Jun;37(6):1049-1057. doi: 10.1111/dme.14289. Epub 2020 Apr 25. PMID 32125000
- [Background] Chen C, Cohrs CM, Stertmann J, Bozsak R, Speier S. Human beta cell mass and function in diabetes: Recent advances in knowledge and technologies to understand disease pathogenesis. Mol Metab. 2017 Jul 8;6(9):943-957. doi: 10.1016/j.molmet.2017.06.019. eCollection 2017 Sep. PMID 28951820
- [Background] Boughton CK, Munro N, Whyte M. Targeting beta-cell preservation in the management of type 2 diabetes. British Journal of Diabetes and Vascular Disease. Published online 2017. doi:10.15277/bjd.2017.148
- [Background] Butler AE, Janson J, Bonner-Weir S, Ritzel R, Rizza RA, Butler PC. Beta-cell deficit and increased beta-cell apoptosis in humans with type 2 diabetes. Diabetes. 2003 Jan;52(1):102-10. doi: 10.2337/diabetes.52.1.102. PMID 12502499
- [Background] Saisho Y. Importance of Beta Cell Function for the Treatment of Type 2 Diabetes. J Clin Med. 2014 Aug 14;3(3):923-43. doi: 10.3390/jcm3030923. PMID 26237486
- [Background] Saisho Y. An emerging new concept for the management of type 2 diabetes with a paradigm shift from the glucose-centric to beta cell-centric concept of diabetes - an Asian perspective. Expert Opin Pharmacother. 2020 Sep;21(13):1565-1578. doi: 10.1080/14656566.2020.1776262. Epub 2020 Jun 10. PMID 32521177
- [Background] RISE Consortium. Lack of Durable Improvements in beta-Cell Function Following Withdrawal of Pharmacological Interventions in Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes. Diabetes Care. 2019 Sep;42(9):1742-1751. doi: 10.2337/dc19-0556. Epub 2019 Jun 9. PMID 31178434
- [Background] Standl E. The importance of beta-cell management in type 2 diabetes. Int J Clin Pract Suppl. 2007 Jun;(153):10-9. doi: 10.1111/j.1742-1241.2007.01360.x. PMID 17594389
- [Background] Kahleova H, Tura A, Hill M, Holubkov R, Barnard ND. A Plant-Based Dietary Intervention Improves Beta-Cell Function and Insulin Resistance in Overweight Adults: A 16-Week Randomized Clinical Trial. Nutrients. 2018 Feb 9;10(2):189. doi: 10.3390/nu10020189. PMID 29425120
- [Background] Zhyzhneuskaya SV, Al-Mrabeh A, Peters C, Barnes A, Aribisala B, Hollingsworth KG, McConnachie A, Sattar N, Lean MEJ, Taylor R. Time Course of Normalization of Functional beta-Cell Capacity in the Diabetes Remission Clinical Trial After Weight Loss in Type 2 Diabetes. Diabetes Care. 2020 Apr;43(4):813-820. doi: 10.2337/dc19-0371. Epub 2020 Feb 14. PMID 32060017
- [Background] Lean MEJ, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Welsh P, Kean S, Ford I, McConnachie A, Messow CM, Sattar N, Taylor R. Durability of a primary care-led weight-management intervention for remission of type 2 diabetes: 2-year results of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 May;7(5):344-355. doi: 10.1016/S2213-8587(19)30068-3. Epub 2019 Mar 6. PMID 30852132
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Davis BC, Jamshed H, Peterson CM, Sabate J, Harris RD, Koratkar R, Spence JW, Kelly JH Jr. An Intensive Lifestyle Intervention to Treat Type 2 Diabetes in the Republic of the Marshall Islands: Protocol for a Randomized Controlled Trial. Front Nutr. 2019 Jun 5;6:79. doi: 10.3389/fnut.2019.00079. eCollection 2019. PMID 31231656
- [Background] Glechner A, Keuchel L, Affengruber L, Titscher V, Sommer I, Matyas N, Wagner G, Kien C, Klerings I, Gartlehner G. Effects of lifestyle changes on adults with prediabetes: A systematic review and meta-analysis. Prim Care Diabetes. 2018 Oct;12(5):393-408. doi: 10.1016/j.pcd.2018.07.003. Epub 2018 Aug 1. PMID 30076075
- [Background] Tonstad S, Stewart K, Oda K, Batech M, Herring RP, Fraser GE. Vegetarian diets and incidence of diabetes in the Adventist Health Study-2. Nutr Metab Cardiovasc Dis. 2013 Apr;23(4):292-9. doi: 10.1016/j.numecd.2011.07.004. Epub 2011 Oct 7. PMID 21983060
- [Background] Abderrahmani A, Niederhauser G, Favre D, Abdelli S, Ferdaoussi M, Yang JY, Regazzi R, Widmann C, Waeber G. Human high-density lipoprotein particles prevent activation of the JNK pathway induced by human oxidised low-density lipoprotein particles in pancreatic beta cells. Diabetologia. 2007 Jun;50(6):1304-14. doi: 10.1007/s00125-007-0642-z. Epub 2007 Apr 17. PMID 17437081
- [Background] Plaisance V, Brajkovic S, Tenenbaum M, Favre D, Ezanno H, Bonnefond A, Bonner C, Gmyr V, Kerr-Conte J, Gauthier BR, Widmann C, Waeber G, Pattou F, Froguel P, Abderrahmani A. Endoplasmic Reticulum Stress Links Oxidative Stress to Impaired Pancreatic Beta-Cell Function Caused by Human Oxidized LDL. PLoS One. 2016 Sep 16;11(9):e0163046. doi: 10.1371/journal.pone.0163046. eCollection 2016. PMID 27636901
- [Background] Lee DH. Lipoproteins and beta-Cell Functions: From Basic to Clinical Data. Diabetes Metab J. 2014 Aug;38(4):274-7. doi: 10.4093/dmj.2014.38.4.274. No abstract available. PMID 25215273
- [Background] Nakhjavani M, Khalilzadeh O, Khajeali L, Esteghamati A, Morteza A, Jamali A, Dadkhahipour S. Serum oxidized-LDL is associated with diabetes duration independent of maintaining optimized levels of LDL-cholesterol. Lipids. 2010 Apr;45(4):321-7. doi: 10.1007/s11745-010-3401-8. Epub 2010 Mar 12. PMID 20224977
- [Background] Wang J, Wang H. Oxidative Stress in Pancreatic Beta Cell Regeneration. Oxid Med Cell Longev. 2017;2017:1930261. doi: 10.1155/2017/1930261. Epub 2017 Aug 3. PMID 28845211
- [Background] Samadi A, Gurlek A, Sendur SN, Karahan S, Akbiyik F, Lay I. Oxysterol species: reliable markers of oxidative stress in diabetes mellitus. J Endocrinol Invest. 2019 Jan;42(1):7-17. doi: 10.1007/s40618-018-0873-5. Epub 2018 Mar 21. PMID 29564756
- [Background] Ferderbar S, Pereira EC, Apolinario E, Bertolami MC, Faludi A, Monte O, Calliari LE, Sales JE, Gagliardi AR, Xavier HT, Abdalla DS. Cholesterol oxides as biomarkers of oxidative stress in type 1 and type 2 diabetes mellitus. Diabetes Metab Res Rev. 2007 Jan;23(1):35-42. doi: 10.1002/dmrr.645. PMID 16634125
- [Background] Maldonado-Pereira L, Schweiss M, Barnaba C, Medina-Meza IG. The role of cholesterol oxidation products in food toxicity. Food Chem Toxicol. 2018 Aug;118:908-939. doi: 10.1016/j.fct.2018.05.059. Epub 2018 Jun 27. PMID 29940280
- [Background] J. V. Vicente S, Sampaio G, Ferrari C, Torres E. Oxidation of Cholesterol in Foods and Its Importance for Human Health. Vol 28.; 2012. doi:10.1080/87559129.2011.594972
- [Background] Lyons MA, Samman S, Gatto L, Brown AJ. Rapid hepatic metabolism of 7-ketocholesterol in vivo: implications for dietary oxysterols. J Lipid Res. 1999 Oct;40(10):1846-57. PMID 10508204
- [Background] Staprans I, Pan XM, Rapp JH, Feingold KR. The role of dietary oxidized cholesterol and oxidized fatty acids in the development of atherosclerosis. Mol Nutr Food Res. 2005 Nov;49(11):1075-82. doi: 10.1002/mnfr.200500063. PMID 16270280
- [Background] Morel DW, Lin CY. Cellular biochemistry of oxysterols derived from the diet or oxidation in vivo. Journal of Nutritional Biochemistry. Published online 1996. doi:10.1016/0955-2863(96)00101-5
- [Background] Linseisen J, Wolfram G. Absorption of cholesterol oxidation products from ordinary foodstuff in humans. Ann Nutr Metab. 1998;42(4):221-30. doi: 10.1159/000012737. PMID 9745108
- [Background] Zmyslowski A, Szterk A. Oxysterols as a biomarker in diseases. Clin Chim Acta. 2019 Apr;491:103-113. doi: 10.1016/j.cca.2019.01.022. Epub 2019 Jan 24. PMID 30685361
- [Background] Endo K, Oyama T, Saiki A, Ban N, Ohira M, Koide N, Murano T, Watanabe H, Nishii M, Miura M, Sekine K, Miyashita Y, Shirai K. Determination of serum 7-ketocholesterol concentrations and their relationships with coronary multiple risks in diabetes mellitus. Diabetes Res Clin Pract. 2008 Apr;80(1):63-8. doi: 10.1016/j.diabres.2007.10.023. Epub 2008 Jan 22. PMID 18207277
- [Background] Indaram M, Ma W, Zhao L, Fariss RN, Rodriguez IR, Wong WT. 7-Ketocholesterol increases retinal microglial migration, activation, and angiogenicity: a potential pathogenic mechanism underlying age-related macular degeneration. Sci Rep. 2015 Mar 16;5:9144. doi: 10.1038/srep09144. PMID 25775051
- [Background] Fu D, Wu M, Zhang J, Du M, Yang S, Hammad SM, Wilson K, Chen J, Lyons TJ. Mechanisms of modified LDL-induced pericyte loss and retinal injury in diabetic retinopathy. Diabetologia. 2012 Nov;55(11):3128-40. doi: 10.1007/s00125-012-2692-0. Epub 2012 Aug 31. PMID 22935961
- [Background] Weigel TK, Kulas JA, Ferris HA. Oxidized cholesterol species as signaling molecules in the brain: diabetes and Alzheimer's disease. Neuronal Signal. 2019 Dec;3(4):NS20190068. doi: 10.1042/NS20190068. Epub 2019 Nov 28. PMID 32269839
- [Background] Odegaard AO, Jacobs DR Jr, Sanchez OA, Goff DC Jr, Reiner AP, Gross MD. Oxidative stress, inflammation, endothelial dysfunction and incidence of type 2 diabetes. Cardiovasc Diabetol. 2016 Mar 24;15:51. doi: 10.1186/s12933-016-0369-6. PMID 27013319
- [Background] Cnop M, Hannaert JC, Grupping AY, Pipeleers DG. Low density lipoprotein can cause death of islet beta-cells by its cellular uptake and oxidative modification. Endocrinology. 2002 Sep;143(9):3449-53. doi: 10.1210/en.2002-220273. PMID 12193557
- [Background] Anderson A, Campo A, Fulton E, Corwin A, Jerome WG 3rd, O'Connor MS. 7-Ketocholesterol in disease and aging. Redox Biol. 2020 Jan;29:101380. doi: 10.1016/j.redox.2019.101380. Epub 2019 Nov 14. PMID 31926618
- [Background] Murakami H, Tamasawa N, Matsui J, Yasujima M, Suda T. Plasma oxysterols and tocopherol in patients with diabetes mellitus and hyperlipidemia. Lipids. 2000 Mar;35(3):333-8. doi: 10.1007/s11745-000-0530-1. PMID 10783011
- [Background] Rodriguez-Estrada MT, Garcia-Llatas G, Lagarda MJ. 7-Ketocholesterol as marker of cholesterol oxidation in model and food systems: when and how. Biochem Biophys Res Commun. 2014 Apr 11;446(3):792-7. doi: 10.1016/j.bbrc.2014.02.098. Epub 2014 Feb 28. PMID 24589732
- [Background] Birlouez-Aragon I, Saavedra G, Tessier FJ, Galinier A, Ait-Ameur L, Lacoste F, Niamba CN, Alt N, Somoza V, Lecerf JM. A diet based on high-heat-treated foods promotes risk factors for diabetes mellitus and cardiovascular diseases. Am J Clin Nutr. 2010 May;91(5):1220-6. doi: 10.3945/ajcn.2009.28737. Epub 2010 Mar 24. PMID 20335546
- [Background] Economic Research Service. Commodity consumption by population characteristics. United States Department of Agriculture. Published 2012. http://www.ers.usda.gov/data-products/commodity-consumption-by-population-characteristics.aspx
- [Background] Kahleova H, Fleeman R, Hlozkova A, Holubkov R, Barnard ND. A plant-based diet in overweight individuals in a 16-week randomized clinical trial: metabolic benefits of plant protein. Nutr Diabetes. 2018 Nov 2;8(1):58. doi: 10.1038/s41387-018-0067-4. PMID 30405108
- [Background] Report NDS. National Diabetes Statistics Report, 2020. National Diabetes Statistics Report. Published online 2020.
- [Background] Lin J, Thompson TJ, Cheng YJ, Zhuo X, Zhang P, Gregg E, Rolka DB. Projection of the future diabetes burden in the United States through 2060. Popul Health Metr. 2018 Jun 15;16(1):9. doi: 10.1186/s12963-018-0166-4. PMID 29903012
- [Background] Mehta SP, Jarvis A, Standifer D, Warnimont C. International physical activity questionnaire. Critical Reviews in Physical and Rehabilitation Medicine. Published online 2018. doi:10.1615/CritRevPhysRehabilMed.2018026180